CLINICAL TRIAL: NCT04117360
Title: Orthognathic Speech Pathology: Phonetic Contrasts of Patients With Dentofacial Discrepancies With Pre- and Post-Treatment Analyses
Brief Title: Orthognathic Speech Pathology: Phonetic Contrasts of Patients With Dental Discrepancies Pre- and Post-Treatment Analyses
Acronym: OSP
Status: Recruiting | Type: Observational
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: North Carolina State University (Other)
Responsible Party: Sponsor
Other Study IDs: 19-1196
Record Dates: First submitted 2019-10-03; First posted 2019-10-07 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Dentofacial Abnormalities; Dentofacial Deformities; Dentofacial Anomalies, Including Malocclusion; Malocclusion; Malocclusion in Children; Dentofacial Disharmony; Skeletal Malocclusion; Skeletal Malformation; Speech Sound Disorder; Speech Disorders
Keywords: Dentofacial Disharmony; Skeletal malocclusion; Speech Sound Disorder; Spectral Moment Analysis; Tongue Ultrasound; Orthognathic Surgery
MeSH Terms: conditions — Dentofacial Deformities; Malocclusion; Speech Sound Disorder; Speech Disorders | interventions — Orthognathic Surgery; Orthodontics

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Dentofacial Disharmony Patients: Dentofacial disharmony patients who are seeking jaw surgery in UNC oral and maxillofacial surgery department and are seen in UNC orthodontic dentofacial disharmony clinic.
  Interventions: Other: Orthognathic surgery and Orthodontics

INTERVENTIONS:
Other: Orthognathic surgery and Orthodontics — This study is observational. All subjects identified to participate will be undergoing orthognathic jaw surgery and orthodontic treatment.

SUMMARY:
The investigators are studying how speech is effected by jaw and tooth position in jaw surgery patients. Eighty percent of our jaw surgery patients have speech pathologies, compared to five percent of the general population, but speech pathologists do not understand why. The investigators hypothesize that open bites and underbites prevent most patients from being able to pronounce words normally and surgical correction will lead to improvement in speech. Patients will be audio recorded speaking and patients' tongue gestures ultrasound recorded before and after their jaw surgeries to observe what changes occur in their speech and tongue movements.

DETAILED DESCRIPTION:
Purpose: The investigators are studying how phoneme distortion is effected by jaw disproportions in dentofacial disharmony (DFD) patients and whether speech improves after orthognathic surgery and orthodontic treatment. Spectral moment and tongue gestural analysis are being used to mechanistically determine how jaw position effects speech. The investigators hypothesize that skeletal open and underbites contribute to phoneme distortion and tongue gestural changes that improve following surgical correction of jaw position. All DFD patients are already seeking treatment from orthodontics and oral surgery. The study will observe how their speech changes before and after treatment. There is no randomization or intervention involved.

Aim 1: Qualify the prevalence of auditory and visual speech distortions in the DFD population. Aim 2: Quantitatively evaluate the first spectral moment (kHz) of four articulating consonant sounds (/t/, /k/, /s/, and /?/ pronounced "sh"). Quantify and analyze the changes in speech distortions for orthognathic patients pre and post-operation. Aim 3: Evaluate tongue posture during speech with patients from Aim 2 pre and post-operation.

Participants:

Participants: Patients of the UNC dentofacial disharmony (DFD) clinic who have undergone orthognathic surgery for correction of jaw disharmonies.

Procedures (methods):

Patients will be recorded pronouncing a series of words highlighting a range of phonetic contrasts including --/s-sh/ and t-k/. words each presented on a screen using PowerPoint, 3 times each with carrier phrases). Recordings include an acoustic feed, a profile video of the jaws plus lips, and ultrasound imaging of the tongue relative to the palate and jaws. Research staff will score audio recordings according to their spectral moments and ultrasound recordings according to tongue movement and associate findings with degree of dental discrepancy. Prospective recordings will be collected at three timepoints: 1-3 months prior to jaw surgery, 3-8 months and 9-15 months post-operation for 60 overbite, 60 openbite and 60 underbite DFD patients. These time points were selected to co-occur with patients' surgical check-ups to ensure reliable data collection while minimizing confounding factors such as severe facial swelling and splint placement which occur immediately after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Jaw surgery patient at UNC with a skeletal open bite, underbite or overjet greater than 5mm.
* Age 15-40 years

Exclusion Criteria:

* Hearing loss
* Learned English as a second language
* Significant regional accent, as characterized by a speech pathologist
* Developmental delay, performing several grade levels below age bracket
* history of craniofacial disorder
* genetic syndrome associated with known craniofacial presentation
* history of craniofacial trauma
* history of prior craniofacial surgery (excluding extractions and dental procedures)
* Jaw surgery without fixed orthodontic appliances

Ages: 15 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The study population includes healthy patients who present in our oral surgery and/or orthodontic dentofacial disharmony clinics with skeletal underbites, open bites, and/or excessive overjet. These patients have decided (prior to our study) to pursue orthodontic treatment combined with orthognathic surgery to address their jaw disproportions.
Sampling Method: Non-Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2019-09-11 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Change in Speech Distortion Phonemes over Time | pre-operation through 9-15 months post-operation
  Audio recordings of consonant phonemes will be quantitatively analyzed using spectral moment analysis yielding mean values.
Change in Quantitative Tongue Gestures over Time | pre-operation through 9-15 months post-operation
  Ultrasound analysis of tongue posture to quantitatively describe tongue position during speech.

CONTACTS AND LOCATIONS:
Overall Officials: Laura A Jacox, PhD, DMD, MS, Principal Investigator — Professor
Locations (1):
- University of North Carolina, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No
Our data includes video, audio and ultrasound recordings. This is not data that can be shared and maintained confidentially while meeting HIPAA guidelines.